CLINICAL TRIAL: NCT02465190
Title: Effectiveness of Trivalent Inactivated Influenza Maternal Vaccination Among Pregnant Women and Their Newborns in South Africa
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Institute for Communicable Diseases, South Africa (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: MatFluVaccSA_v2_11/03/2015
Record Dates: First submitted 2015-04-28; First posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Influenza Viral Infections
Keywords: Vaccine; Effectiveness; Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Nasopharyngeal swabs and aspirates
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a case-control study embedded in a surveillance system to determine the effectiveness of antenatal maternal influenza vaccination against laboratory-confirmed influenza-associated hospitalised illness in infants <6 months of age.

DETAILED DESCRIPTION:
Study design Investigators will conduct a vaccination campaign amongst pregnant women in different areas of South Africa and monitor the effectiveness of the programme. Investigators will then use an unmatched case-control study design.

Vaccination campaigns will be conducted in clinics with active promotion of influenza vaccination. Posters will be placed in clinics recommending influenza vaccination for pregnant women and health education material will be provided. Vaccines will be administered by clinic staff through routine services as vaccination is the recommended standard of care. Dedicated study staff (research assistants) will be placed in each clinic offering vaccination. These staff will assist clinic staff with management of influenza vaccine supplies and documentation of influenza vaccination status in patient records. Vaccination status will be documented in the mother's antenatal records. Investigators will visit all the facilities in the area serving the surveillance hospital and conduct staff training in the facilities where babies are delivered to enter maternal influenza immunization status on the child's vaccination card at the time of administration of the birth dose of polio vaccine.

Identification and enrolment of cases and controls for the estimation of VE against laboratory-confirmed influenza-associated hospitalised illness in infants<6 months of age overall and by HIV status Cases and controls will be identified through active sentinel surveillance for hospitalised medical illness of any diagnosis amongst children aged <6 months. Hospitals where surveillance will be conducted will be large hospitals serving the communities in which the antenatal TIV campaign will be conducted. Investigators will conduct ongoing active surveillance with consecutive patient selection until the required sample size is reached.

Identification and enrolment of cases for monitoring adverse events Dedicated study staff will conduct an information session with women selected for enrolment. These women will be asked for written informed consent prior to participation and non-participation will not affect a woman's eligibility to receive vaccine. Following vaccination administered by the nurse, as per the Department of Health schedule, demographic information, medical history, obstetric history and contact details will be collected from each participant by structured interview. Immediate reactions to the vaccine will be recorded at the time of interview. A separate aide de memoire diary will then be given to each participant. This diary will assist the women to record symptoms experienced in the seven days following vaccination. The symptoms listed will be based on standard collection tool.

Data collection Hospitalised children <6 months For hospitalised children <6 months of age, epidemiologic data will be collected from a parent or caregiver interview, if possible, as well as review of medical and vaccination records of mother (antenatal cards, maternal in-patient cards and antenatal clinic registers) and baby (Road-to-Health cards and clinic registers). Information gathered will include: demographics of mother and baby (age, sex, race), medical history of baby (premature birth, congenital illnesses such congenital heart or lung disease, immunosuppressive or other chronic illness), recent infections, recent antimicrobial use, household characteristics (residence type and number of rooms, number of persons and their ages, questions related to socioeconomic status, exposure to tobacco smoke and indoor air pollution), child-care centre attendance, breast feeding and vaccination history. It will also request educational level of the parent or guardian and if adults or other children in the household had received pneumococcal or influenza vaccines. Information on HIV status will include whether the mother was tested for HIV during pregnancy and her HIV status if tested, whether the patient has been previously tested for HIV and results of such tests, history of underlying illness and previous HIV-associated diagnosis. Nutritional status of the child will be evaluated measuring weight (in kilograms) and length (in centimetres) at the time of admission. If the parent or guardian has a written vaccination record for the case or control child, names, batch numbers and dates of vaccines will be recorded (see determination of vaccination status below). For issues that may change with time (e.g. exposure to cigarette smoke, breastfeeding, day-care attendance), the questions will focus on the 4 weeks (as in 30 or 31 days) before illness.

Adverse birth outcomes For the effectiveness against adverse birth outcomes (prematurity, LBW and SGA) epidemiologic data will primarily be collected from birth records and maternal antenatal records. Information gathered will include: demographics of mother and baby (age (of mother), sex, race), household characteristics (residence type and number of rooms, number of persons and their ages, questions related to socioeconomic status. It will also request educational level of the parent or guardian. Information on HIV status will include whether the mother was tested for HIV during pregnancy and her HIV status if tested. The baby's birthweight and gestational age will be evaluated from delivery and antenatal records. Birthweight (in kilograms) and length (in centimetres) will be documented.

Hospitalised pregnant women and postpartum women, ≥18 years Epidemiologic, clinical presentation, laboratory data as well as information on hospital course will be collected from enrolled patients. A case investigation form will be completed by structured interview. Information gathered will include: demographics (age, sex, race), presenting symptoms, medical history (lung disease, immunosuppressive or other chronic illness including cardiac diseases, chronic renal diseases, diabetes mellitus and similar metabolic disorders), previous hospital admissions, recent infections, recent antimicrobial use, household characteristics (residence type and number of rooms, number of persons and their ages, questions related to socioeconomic status, exposure to tobacco smoke and indoor air pollution) and data on current and previous influenza vaccination. Information on HIV status will include current HIV status and whether the patient has been previously tested for HIV and results of such tests, previous HIV-associated diagnosis, HIV staging. Obesity evaluated measuring weight (in kilograms) and length (in centimetres) at the time of admission. Medical records will be reviewed for inpatient management (antimicrobial use, influenza antiviral therapy and results of investigations conducted) and outcome (admission to ICU, discharged or died).

Monitoring adverse events The diary will be taken home by the participant. Telephone contact will be made with the participant by a study staff member on day eight (or day 7, 9 or 10 if day 8 falls over a weekend) and the contents of the diary will be recovered telephonically. If the study staff are not able to contact the participant on the first attempt, three further documented attempts will be made to contact the patient. Participants will also be request to return their diaries at their next clinic visit. Participating women will be asked to contact the study team if she is hospitalized for any reason in the seven days post-vaccination. A member of the study team will visit the woman in hospital and, using a predesigned form, collect data on the reason for hospitalization.

Logs recording the enrolled patients with their contact details will be kept at each site. Completed data collection forms will be returned to the data centre at NICD for data capture and storage.

ELIGIBILITY:
Inclusion Criteria:

* Cases and controls will meet the following inclusion criteria:

  1. Child admitted to the medical wards at designated surveillance hospitals aged <6 months on day of hospital admission
  2. Mother was eligible to receive influenza vaccination during pregnancy (i.e. pregnant from ~April onwards but actual date will be determined based on actual campaign dates and resident in the area where vaccination was offered)
  3. Nasopharyngeal aspirate collected and influenza rRT-PCR result available
  4. Documented HIV and HIV-exposure status or consent to child and maternal HIV testing (for the endpoint of HIV-status specific VE only)
  5. Consent to inclusion in the study

Study enrolment will occur as follows. Study nurses will review all hospital admissions (paediatric medical and sleep over wards) to study hospitals each day to identify any children meeting study case definitions. Parents or guardians of eligible patients will be approached for enrolment into the case-control study. Parents or guardians will be asked if study staff can collect a nasopharyngeal aspirate specimen from the child. In addition, they will be asked to participate in an interview consisting of a list of standardised questions. Additional information will be obtained from hospital records. If not already tested for HIV by the ward doctors, HIV testing with pre- and post-test counselling will be offered to children and mothers to determine child's HIV and HIV-exposure status.

A register of all patients approached for enrolment but declining study inclusion and reasons for non-enrolment will be complied.

Identification and enrolment of cases and controls for the estimation of VE against adverse birth outcomes (prematurity, LBW, SGA and stillbirth)

Study staff will review all children born at hospitals with maternity wards described in section 9.2 (Study setting and Population 2nd last paragraph) during and up to three months after the influenza season (from May to December each year). Cases and controls will meet the following inclusion criteria:

1. Child born at designated surveillance hospitals
2. Mother was eligible to receive influenza vaccination during pregnancy (i.e pregnant from ~April onwards but actual date will be determined based on actual campaign dates and resident in the area where vaccination was offered)
3. Data on birth outcomes (preterm birth, LBW and SGA) available
4. Documented evidence of maternal TIV vaccination status able to be ascertained
5. Documented HIV and HIV-exposure status or consent to child and maternal HIV testing (for the endpoint of HIV-status specific VE only)
6. Consent to inclusion in the study

Study staff will review all babies born at each hospital each day. Gestational age will be ascertained based on dates using the Ballard system. If the investigators have sufficient data, investigators will explore different cut-off gestational age values for the analysis of preterm birth.

Exclusion Criteria:

- Hospitalised children <6 months

* Children whose mothers were not resident in the area where vaccination was offered during the period of the vaccination campaign.
* Previous inclusion as a case or control Adverse birth outcomes
* Babies with unavailable data on birth outcomes.
* Children whose mothers were not resident in the area where vaccination was offered during the period of the vaccination campaign.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted in Gauteng Province and Western Cape Province in South Africa. Both are urban areas with good access to hospital care for mothers and infants. Babies born to women who were eligible to receive influenza vaccination during pregnancy (i.e. pregnant from April onwards but actual date will be determined based on actual campaign dates and resident in the area where vaccination was offered) will be the study population. Investigators will conduct surveillance for hospitalisations amongst infants <6 months of age. Investigators will conduct surveillance for adverse birth outcomes at identified hospitals. Investigators will conduct surveillance for LRTI hospitalisations among pregnant and postpartum women.
Sampling Method: Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Laboratory-confirmed influenza-associated hospitalised illness in infants<6 months of age | hospitalised infants up to 6 months of age, whose mothers were eligible to have received influenza vaccination and born between March and August.

SECONDARY OUTCOMES:
Laboratory-confirmed influenza-associated hospitalised illness in infants<6 months of age by HIV exposure status | hospitalised infants up to 6 months of age, whose mothers were eligible to have received influenza vaccination and born between March and August.
Laboratory-confirmed influenza-associated hospitalised illness in pregnant women | Pregnant woman admitted to the obstetric or gynaecology wards with cardio-respiratory illness and eligible to have received influenza vaccination for up to 42 days postpartum
Laboratory-confirmed influenza-associated hospitalised illness in post-partum women | up to 42 days postpartum woman admitted to the obstetric or gynaecology wards with cardio-respiratory illness and eligible to have received influenza vaccination.
Occurrence and severity of adverse events following immunization with seasonal influenza vaccine in pregnant women | Pregnant woman admitted to the obstetric or gynaecology wards with cardio-respiratory illness and eligible to have received influenza vaccination for up to 42 days postpartum
Low birth weight | hospitalised infants up to 6 months of age, whose mothers were eligible to have received influenza vaccination and born between March and August.
Preterm birth as determined by gestational age | hospitalised infants up to 6 months of age, whose mothers were eligible to have received influenza vaccination and born between March and August.
Stillbirth | Birth
Small for gestational age birth as determined by birth weight | hospitalised infants up to 6 months of age, whose mothers were eligible to have received influenza vaccination and born between March and August.

CONTACTS AND LOCATIONS:
Overall Officials: Shabir Madhi, PhD, Principal Investigator — National Institute for Communicable Diseases
Locations (1):
- Chris Hani Baragwanath Academic Hospital and National Institute for Communicable Diseases, Johannesburg, Gauteng, South Africa

REFERENCES:
- [Derived] Omer SB, Clark DR, Madhi SA, Tapia MD, Nunes MC, Cutland CL, Simoes EAF, Aqil AR, Katz J, Tielsch JM, Steinhoff MC, Wairagkar N; BMGF Supported Maternal Influenza Immunization Trials Investigators Group. Efficacy, duration of protection, birth outcomes, and infant growth associated with influenza vaccination in pregnancy: a pooled analysis of three randomised controlled trials. Lancet Respir Med. 2020 Jun;8(6):597-608. doi: 10.1016/S2213-2600(19)30479-5. PMID 32526188
- [Derived] Clark DR, Omer SB, Tapia MD, Nunes MC, Cutland CL, Tielsch JM, Wairagkar N, Madhi SA; for BMGF Supported Maternal Influenza Immunization Trials Investigators Group. Influenza or Meningococcal Immunization During Pregnancy and Mortality in Women and Infants: A Pooled Analysis of Randomized Controlled Trials. Pediatr Infect Dis J. 2020 Jul;39(7):641-644. doi: 10.1097/INF.0000000000002629. PMID 32379201
- [Derived] Omer SB, Clark DR, Aqil AR, Tapia MD, Nunes MC, Kozuki N, Steinhoff MC, Madhi SA, Wairagkar N; for BMGF Supported Maternal Influenza Immunization Trials Investigators Group. Maternal Influenza Immunization and Prevention of Severe Clinical Pneumonia in Young Infants: Analysis of Randomized Controlled Trials Conducted in Nepal, Mali and South Africa. Pediatr Infect Dis J. 2018 May;37(5):436-440. doi: 10.1097/INF.0000000000001914. PMID 29443825